CLINICAL TRIAL: NCT04377893
Title: Applying Eye-Gaze Assistive Technology in Daily Life for Children and Youth With Severe Physical Disabilities and Complex Communication Needs
Brief Title: Applying Eye-Gaze Assistive Technology for Children and Youth With Complex Needs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yu-Hsin Hsieh (Other)
Collaborators: Chang Gung University (Other); Jonkoping University (Other); Folke Bernadotte Stiftelsen (Unknown); Stiftelsen Kempe-Carlgrenska Fonden (Unknown); Stiftelsen Clas Groschinskys Minnesfond (Unknown); Helge Ax:son Johnsons Stiftelse (Unknown)
Responsible Party: Sponsor-Investigator, Yu-Hsin Hsieh, Sponsor-Investigator, Stockholm University
Organization: Stockholm University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CGUSU180116
Record Dates: First submitted 2020-04-22; First posted 2020-05-07 (Actual); Last update posted 2021-09-27 (Actual); Status verified 2021-09

CONDITIONS: Self-Help Devices; Eye-Gaze Technology; Severe Physical Disabilities; Communication Disorders
Keywords: Eye-Gaze Assistive Technology; Severe Physical Disabilities; Communication difficulties
MeSH Terms: conditions — Communication Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment arm (Experimental): Participants will receive eye-gaze AT intervention
  Interventions: Device: Eye gaze AT intervention

INTERVENTIONS:
Device: Eye gaze AT intervention — The eye-gaze AT intervention includes eye-gaze AT and service delivery to support the participants using this technology in daily life. The Tobii PCEye Mini (Tobii, Danderyd, Sweden) and specialized software are applied with adaptation to meet each child's individual needs.
  To ensure the consistency of service delivery, two-day courses are conducted before the intervention. The participant's teachers or parents are invited as the main interventionist to facilitate the child's usage of eye-gaze AT in daily life under team support. The service delivery involves parents in joint goal-setting, planning, and jointly review the progress of the usage of eye-gaze AT as a family-centered practice. Individual meetings and individual supports are provided during intervention periods. The collaborative team will perform biweekly follow-up contacts during intervention periods.
  The researcher will conduct the fidelity checklist every month to determine the extent of treatment integrity.

SUMMARY:
The purpose of this research is to investigate the impacts of applying eye-gaze assistive technology (AT) in children and youth with severe disabilities and complex needs in Taiwan, where eye-gaze AT has not been researched for children yet.

DETAILED DESCRIPTION:
Background. Children and youth with severe physical disabilities often have concomitant mental impairments and complex needs in communication, and in building relationships with others. The impairments limit their participation and independence in family, school and community life. By using their eyes, the only movements they can control voluntarily, they may increase communication. Relevant research has shown that using eye-gaze AT was feasible for children with severe physical disabilities to make choices, communicate, interact or perform school tasks despite different learning curves. Use of technology may increase opportunities for engagement and self-determination for children and youth with physical disabilities and complex communication needs in family context or in school, but the research is relatively limited. It still needs more studies across countries and long-term follow-up to investigate the effects of the use of eye-gazed AT in life.

Study Aims. There are two aims in this proposed research. Aim 1: To investigate the preliminary effects of eye-gazed AT for daily participation in daily living for children and youth with severe physical disabilities and communication difficulties in Taiwan.

Aim 2: To investigate the adherence of eye-gazed AT intervention for children and youth with severe physical disabilities and communication difficulties, and the caregivers' satisfaction regarding support children and youth to use eye-gazed AT in daily living in Taiwan.

Methods. This study is conducted as a single subject design with multiple baselines across individuals. The inclusions are non-concurrent and the baselines before the intervention started were randomized with unequal of 14-30 days.

This study enrolls participants from Northern Taiwan. The researcher team contacts the practitioners in hospitals, schools or development centers to assist recruitment.

Study procedure. The eye-gaze AT intervention will be conducted for six months and follow up to seven months since provision. Before the intervention started, each of the five participants is randomly assigned to one of the pre-determined baseline lengths (14-30 days).

Repeated measures were conducted in baseline period with a minimum of five data points to judge the stability of the child's abilities and in intervention phase to establish data trends in the levels of two dependent variables, computer usage in daily living (measured by computer use diary along with log data of FocusMe program (FocusMe Inc., London, UK)), and children's activity performance using eye-gaze AT (performance scale of Canadian Occupational Performance Measure (COPM) rated by the parent or teacher). Systematic manipulation of the independent variable, the eye-gaze AT intervention was introduced in the intervention phase. The process was replicated for at least five participants to demonstrate the experiment-control effects.

In addition, other outcomes related to Activity and Participation, Body Functions and Structures and Environmental dimensions based on ICF-CY framework will be collected at baseline, after the 3-month intervention, after the 6-month intervention and 7-month after provision.

Statistical analysis. The visual analysis of single-case data will be used to determine whether there will be a relationship between the independent and dependent variables. The data of continuous variables will be presented as graphs to visually inspected regarding change of data pattern across phases separately.

Due to the small sample size, descriptive statistics will be used to summarize the results of outcome measures and reported using the narrative summary. For COPM, the score change of more than two points is considered clinically signiﬁcant improvement on both performance and satisfaction scale. Besides, achieving the expected level (0) on a GAS goal is considered successful goal attainment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with severe physical disability without speaking abilities or with communication difficulties (level III~V on the Communication Function Classification System (CFCS); level IV~V on the Gross Motor Function Classification System (GMFCS) and Manual Ability Classification System (MACS);
* Children have intentions to communicate using body movement, sounds, facial expressions or others, measured by Communication Matrix (Rowland, 2010) with some emerging skills in level 3;
* No or limited possibilities to interact with computers using an input method other than EGAT (e.g. switch or touchpads)
* With access to eye-gazed AT but not used it in daily routines; if possible, new to eye-gaze AT;
* The parent or the teacher agrees to participate in supporting children to use eye-gaze AT in everyday life during the research period;
* The therapist who has worked with the child demonstrated motivation to participate in this intervention.

Exclusion Criteria:

* Progressive diseases that caused functional declines, or serious illness

Ages: 1 Year to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Actual)
Dates: Start 2019-09-19 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
The Computer Use Diary | is collected everyday for 8 months.
  to measure the children´s computer usage in daily living throughout the research period. Parents and teachers observe and document the computer use at home, school and/or center, including duration of use for each activity and type and number of computer activities per day. To increase the reliability of using documentation data from parents or teachers, we will compare with log data from the FocusMe program (FocusMe Inc., London, UK) which monitors the duration and types of app/software the children use eye-gaze AT each time to enhance internal validity.
Changes of Canadian Occupational Performance Measure (COPM) | The performance of COPM is monitored twice a week using the proxy ratings by parent or the teacher for 8 months. The satisfaction of COPM is measured at baseline, 3 months and 6 months since intervention provision.
  to interview the parents or teachers to prioritize goals for daily participation activities using an eye-gazed AT and rate the level of children's performance and satisfaction of children's performance using a 10-point scale (1-10). Higher scores means better performance or higher satisfaction on children's performance.
Changes of Goal Attainment Scaling (GAS) | is collected at 3 months and 6 months since intervention provision.
  to evaluate the goals of meaningful use in school and at home with eye-gazed AT. The instrument has five levels of scale values from -2 (starting level) to +2 (more than expected)

SECONDARY OUTCOMES:
Communication Matrix | is measured at baseline, 3 months and 6 months since intervention provision.
  to evaluate the communicative functions for early communication behaviors through a telephone or face to face interview with proxy persons.
Chinese version of Psychosocial Impact of Assistive Devices Scale (PIADS-C) | is measured at baseline (if the child uses other AT for communication) and after 6-month intervention.
  is used to assess the impact of AT on the subjective well-being of end users by proxy persons, including three subscales of competence, adaptability and self-esteem. Each subscale score ranges from -3 to +3, and higher scores indicate better outcomes.
KIDSCREEN-10 parent version | is measured at baseline and after 6-month intervention.
  to evaluate child´s physical, psychological and social well-being. Items are answered on a 5-point Likert-type scale and responses are summed and transformed into T-score with a mean of 50 and a standard deviation of approximately 10. A high score is indicative of a better health-related quality of life.
The Taiwanese Version of Quebec User Evaluation of Satisfaction with Assistive Technology (T- QUEST) | is measured after 6-month intervention.
  to evaluate parents' and teachers' satisfaction with the eye-gazed AT as an assistive device and with the service provided related to the eye-gazed AT. Each item ranges from 1 "Not satisfied at all" to 5 "Very satisfied." Higher values represent higher satisfaction.
COMPASS Aim test | Five trials with 12 targets in each trial will be conducted at baseline, 3 months and 6 months since intervention provision.
  to measure the eye gaze performance (time on task and accuracy) with the eye-gazed AT.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Special Education, Stockholm University, Stockholm, Sverige, Sweden

IPD SHARING:
Plan to Share IPD: No